CLINICAL TRIAL: NCT06292897
Title: Integrating Tissue-based Spatial Information to Elucidate How Obesity-induced Tumour Metabolites Drive Prostate Cancer Progression
Brief Title: Using Tissue-based Spatial Data to Understand How Obesity-related Tumor Metabolites Fuel Prostate Cancer Progression
Acronym: OBESITA'&PCa
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: National Research Council (Unknown)
Responsible Party: Principal Investigator, Giancarlo Albo, associate professor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 3312
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostate Neoplasm; Prostatic Neoplasm; Obesity
MeSH Terms: conditions — Prostatic Neoplasms; Obesity | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese individuals [Body Mass Index (BMI) > 30 affected by prostate cancer
  Interventions: Other: observational study
- normal-weight individuals [18 < BMI < 25] affected by prostate cancer

INTERVENTIONS:
Other: observational study — observational study
  Groups: obese individuals [Body Mass Index (BMI) > 30 affected by prostate cancer

SUMMARY:
Evaluate the protein expression of lactate dehydrogenase enzyme (LDHA) and MCT-1/-4 transporters, involved in lactate synthesis and transport, in prostate carcinoma tissues from severely overweight/obese (BMI > 27.5) and non-severely overweight/normoweight (BMI < 27.5) patients affected by prostate carcinoma.

ii. Characterize the immune infiltrate in the prostate carcinoma of the aforementioned patients.

iii. Assess the association between intra-tumoral lactate accumulation (using LDHA and MCT-4 protein expression levels as readouts) and alterations in the tumor immune microenvironment and/or deregulation of relevant oncogenic pathways.

ELIGIBILITY:
Inclusion Criteria:

* affected by prostate cancer

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients affected bt prostate cancer both obese or not obese
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Assess the protein expression of LDHA enzyme and MCT-1/-4 transporters in prostate carcinoma | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Cà Granda Ospedale Maggiore Policlinico Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided